CLINICAL TRIAL: NCT06837454
Title: French Prospective Observational Study in Patients Eligible for Systemic Therapy for Atopic Dermatitis (AD)
Acronym: FRAME
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17667; U1111-1279-3382 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-01-28; First posted 2025-02-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atopic Dermatitis: The study plans to collect information on patients during visits according to clinical practice. Enrolled patients will receive AD treatment of marketed drugs prescribed by the specialty physician. No investigational drug will be given for the purpose of this study.

SUMMARY:
The objective of the study is to describe the therapeutic management of patients more than or equal to 18 years old eligible for systemic therapy or treated by systemic therapy for atopic dermatitis (AD). This study will be proposed to a sample of French dermatologists experienced in the management of AD, practicing in hospital centers and/or office-based dermatologists. The study will be conducted in real conditions of practice, systemic treatment decisions will be taken at the sole initiative of the participating physician irrespective of the patient enrollment decision. Each patient will be followed-up in routine care setting for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Patient with moderate to severe AD according to the Investigator's judgment and

  1. Patient eligible to systemic treatment as Atopic Dermatitis Control Tool (ADCT) more than or equal to (≥) 7 and/or use topical corticosteroids (TCS) more than (>) 90 gram (g)/month and/or TCS are not advisable.

     or
  2. Patient currently under systemic treatment.
* Able to understand and complete study-related questionnaires.

Exclusion Criteria:

* Any condition that, in the opinion of the Investigator, may interfere with patient's ability to participate in the study, such as short life expectancy, substance abuse, severe cognitive impairment, or other comorbidities that can predictably prevent the patient from adequately completing, as per routine care, the schedule of visits and assessments
* Patient receiving systemic therapy only for a disease other than AD.
* Patient participating in any interventional clinical trial at the time of enrolment.
* Patient is under tutorship or curatorship; patient under safeguard of justice or deprived of his/her liberty by an administrative or court decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating in this study will be more than equal to (≥) 18 years old, managed in France for moderate to severe AD, and who are either eligible to systemic treatment or currently under systemic treatment, in realworldsettings within the inclusion period.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-05-13 (Estimated); Study Completion 2027-05-13 (Estimated)

PRIMARY OUTCOMES:
Previous and Current Treatments for Atopic Dermatitis (AD) | Baseline, month 6 and month 12
  List of previous and current treatments for AD based on physician-reported data will be assessed.
Atopic Comorbidities: Previous and Current Therapeutic Management | Baseline, month 6 and month 12
  Description of previous and current therapeutic management of atopic comorbidities over time based on physician-reported data will be assessed.
Change from Baseline in Drug Survival for Systemic Treatments for AD by Name and Dose | Baseline, month 6 and month 12
  Drug survival is defined as the time from the start of treatment to the end or discontinuation of treatment with no changes. If a patient has multiple drug survival events for the same treatment, the longest drug survival will be used in the data summarization. The drug survival will be illustrated using a Kaplan-Meier plot.
Compliance for AD Treatments | Baseline, month 6 and month 12
  Compliance for AD treatments will be assessed by the physician.

SECONDARY OUTCOMES:
Demographic Characteristics of Participants | Baseline
  Demographics characteristics including birth date, gender, and socio-professional category, height, weight, phototype (type I to type VI according to Fitzpatrick's classification).
Medical History and AD history | Baseline
  Medical history will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA) codes of System Organ Class (SOC) and Preferred Terms (PT).
Change from Baseline in AD Severity | Baseline, month 6 and month 12
  Change from baseline in AD severity assessed through physician-reported persistence with prescribed therapy.
Atopic Comorbidities | Baseline, month 6 and month 12
  Description of the presence, evolution, and therapeutic management of atopic comorbidities over time based on physician-reported data.
Non-atopic Comorbidities | Baseline, month 6 and month 12
  Description of the presence, evolution, and therapeutic management of non-atopic comorbidities over time based on physician-reported data.
Use of Psychoactive Substances | Baseline, month 6 and month 12
  Description of the use of psychoactive substances over time based on patient-reported data.
Change from Baseline in Itch Assessment | Baseline, month 6 and month 12
  Itch assessment (Worst-Itch Numeric Rating Scale, WI-NRS) will be rated from 0 to 10 on average during the past 7 days, completed by the observing physician after questioning of patient; 0 = no itch and 10 = the worst imaginable itch.
Change from Baseline in Sleep Disturbance NRS | Baseline, month 6 and month 12
  NRS sleep disturbance will be rated from 0 to 10 on average during the past 7 days, completed by the observing physician after questioning of patient; 0 = "sleep not disturbed at all" (best possible sleep) and 10 = "sleep extremely disturbed (worst possible sleep)".
Change from Baseline in Skin Pain NRS | Baseline, month 6 and month 12
  Skin pain NRS will be rated from 0 to 10 on average during the past 7 days prior to the visit. On a scale of 0 to 10, with 0 being 'no skin pain at all' and 10 being 'the worst imaginable skin pain'.
Change from Baseline in AD Disease Control Using the Atopic Dermatitis Control Tool (ADCT) | Baseline, month 6 and month 12
  ADCT is a questionnaire to assess patient-self-perceived control of their AD with a total score from 0 to 24; higher scores indicate lower AD control.
Change from Baseline in Dermatology Life Quality Index (DLQI) | Baseline, month 6 and month 12
  DLQI is a 10-item questionnaire to measure dermatology specific quality of life (QoL). DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
Change from Baseline in Psychological Comorbidities Assessed using Hospital Anxiety and Depression Scale (HADS) | Baseline, month 6 and month 12
  The HADS is a 14-item patient-reported outcomes measure used to assess states of anxiety and depression over the past week. It is comprised of 7 items assessing anxiety and depression respectively. A Total score is out of 42 (21 per subscale). Higher scores indicate greater levels of anxiety and/or depression.
Cumulative Life Course Impairment (CLCI) - for Physicians in Hospital Centers | Baseline, month 6 and month 12
  CLCI-r instrument determines retrospectively which changes and effects the patients have already experienced due to the disease over their entire disease course.
  CLCI-p determines the patient's current situation and thus identifies risk areas in which the patient could experience burdens in the future.
Change from Baseline in Patient's Treatment Satisfaction Score Using the Patient Global Assessment of Treatment Effect (PGATE) | Baseline, month 6 and month 12
  Patient's treatment satisfaction score will be assessed using Patient Global Assessment of Treatment Effect (PGATE). PGATE is an assessment tool used to rate the treatment effect of the medication on atopic dermatitis (AD), with scores ranging from 0 to 4 (0 = poor; 1 = fair; 2 = good; 3 = very good; 4 = excellent), i.e., higher score indicated higher treatment effect.
Evolution of Atopic Comorbidities | Baseline, month 6 and month 12
  Evolution of atopic comorbidities over time, assessed through physician-reported status, occurrence of new diagnoses and persistence of existing conditions.
Management of AD from First Diagnosis | Baseline, month 6 and month 12
  History of healthcare pathway of participant related to AD will be assessed by the physician (if participant had appointment with other healthcare provider for AD).
Therapeutic Education | Baseline, month 6 and month 12
  History of healthcare pathway of participant related to AD will be assessed by the physician (if participant received therapeutic education).
Cost of Emollients and Hygiene Products | At month 12
  Cost of emollients, hygiene products etc. during the last month of the study visit will be assessed.
Sick Leaves Related to AD | Baseline, month 6 and month 12
  Number of sick leaves participant has taken related to AD since the last visit or over the last 6 months.
Hospitalization with Overnight Stay Related to AD | Baseline, month 6 and month 12
  Overnight hospitalization related to AD since the last visit or over the last 6 months.

CONTACTS AND LOCATIONS:
Locations (56):
- France (56):
  - Investigational Site Number: 2500051, Aix-en-Provence
  - Investigational Site Number: 2500023, Amiens
  - Investigational Site Number: 2500004, Angers
  - Investigational Site Number: 2500017, Angers
  - Investigational Site Number: 2500050, Arès
  - Investigational Site Number: 2500063, Arès
  - Investigational Site Number: 2500054, Bayonne
  - Investigational Site Number: 2500043, Bezannes
  - Investigational Site Number: 2500040, Biarritz
  - Investigational Site Number: 2500036, Bordeaux
  - Investigational Site Number: 2500053, Bordeaux
  - Investigational Site Number: 2500013, Chalon-sur-Saône
  - Investigational Site Number: 2500026, Chalon-sur-Saône
  - Investigational Site Number: 2500046, Chalon-sur-Saône
  - Investigational Site Number: 2500041, Châlons-en-Champagne
  - Investigational Site Number: 2500018, Cherbourg
  - Investigational Site Number: 2500020, Cholet
  - Investigational Site Number: 2500048, Clermond Ferrand
  - Investigational Site Number: 2500059, Contamine-sur-Arve
  - Investigational Site Number: 2500010, Dunkirk
  - Investigational Site Number: 2500049, Fort-de-france
  - Investigational Site Number: 2500032, La Ravoire
  - Investigational Site Number: 2500044, La Ravoire
  - Investigational Site Number: 2500011, La Roche-sur-Yon
  - Investigational Site Number: 2500037, La Tronche
  - Investigational Site Number: 2500056, Le Mans
  - Investigational Site Number: 2500068, Le Mans
  - Investigational Site Number: 2500001, Le Mans
  - Investigational Site Number: 2500012, Le Puy-en-Velay
  - Investigational Site Number: 2500003, Limoges
  - Investigational Site Number: 2500031, Loperhet
  - Investigational Site Number: 2500060, Marseille
  - Investigational Site Number: 2500055, Monaco
  - Investigational Site Number: 2500058, Mont-de-Marsan
  - Investigational Site Number: 2500033, Niort
  - Investigational Site Number: 2500005, Paris
  - Investigational Site Number: 2500030, Paris
  - Investigational Site Number: 2500009, Paris
  - Investigational Site Number: 2500028, Périgueux
  - Investigational Site Number: 2500027, Périgueux
  - Investigational Site Number: 2500029, Rennes
  - Investigational Site Number: 2500035, Rennes
  - Investigational Site Number: 2500021, Romans-sur-Isère
  - Investigational Site Number: 2500022, Rouen
  - Investigational Site Number: 2500025, Saint-Etienne
  - Investigational Site Number: 2500062, Saint-Gervais-les-Bains
  - Investigational Site Number: 2500034, Saint-Maur-des-Fossés
  - Investigational Site Number: 2500008, Saint-Maur-dès-Faussés
  - Investigational Site Number: 2500045, Saint-Quentin
  - Investigational Site Number: 2500019, Sainte-Maxime
  - Investigational Site Number: 2500015, Toulouse
  - Investigational Site Number: 2500016, Tours
  - Investigational Site Number: 2500038, Vannes
  - Investigational Site Number: 2500024, Villefranche-sur-Saône
  - Investigational Site Number: 2500052, Villeurbanne
  - Investigational Site Number: 2500066, Villeurbanne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org